CLINICAL TRIAL: NCT01093482
Title: Third Prospective, Observational, International, Multicenter Study on Mechanical Ventilation
Brief Title: Third International Study on Mechanical Ventilation
Acronym: ISMV
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Principal Investigator, Andres Esteban, MD, Hospital Universitario Getafe
Other Study IDs: ISMV-2010
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Results first posted 2018-01-26 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Acute Respiratory Failure
Keywords: mechanical ventilation; epidemiology; outcomes; mortality; weaning; sedation; non-invasive positive pressure ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mechanically ventilated patients: 1. Patients who are admitted to the participating intensive care units and require invasive mechanical ventilation (endotracheal tube or tracheostomy) for more than 12 hours.
  2. Patients who are admitted to the participating intensive care units and require non-invasive mechanical ventilation (Bilevel positive airway pressure (BIPAP) or continuous positive airway pressure (CPAP) with nasal or facial mask) for more than 1 hour.

SUMMARY:
The objective of this study is to obtain a better understanding of the spectrum of use of mechanical ventilation in intensive care units:

1. Main analysis: To know the all-cause mortality rate in mechanically ventilated patients
2. Secondary analyses:

   * To know the current status of mechanical ventilation in the intensive care unit and determine the number and percentage of patients who are admitted to an intensive care unit and require mechanical ventilation.
   * To compare the results with prior data collected in previous observational studies (1998 and 2004)
   * Non-invasive positive pressure ventilation
   * Weaning
   * Use of adjuvant therapies as steroids or selective digestive decontamination
   * Sedation including prevalence of delirium in mechanically ventilated patients
   * Prediction of the duration of mechanical ventilation
   * Other

DETAILED DESCRIPTION:
Mechanical ventilation is commonly used in patients admitted to intensive care units. Clinical studies have investigated some of the aspects associated with its utilization, and have contributed to improve the knowledge and management of patients with acute respiratory failure. In 1998 the invesgtigators conducted the first international study on mechanical ventilation, including 5183 patients who were mechanically ventilated longer than 12 hours (Esteban A. JAMA 2002). Six years later, the investigators carried out the second international study on mechanical ventilation including 4968 patients. These studies allowed us to analyze the evolution of mechanical ventilation and to judge the concordance of practice with results of randomized trials (Esteban A. Am J Respir Crit Care 2008). The main finding of this study was the high degree of concordance between observed changes in mechanical ventilation practice and changes predicted from reports of randomized controlled trials. However, despite apparently beneficial changes in ventilatory practice, the investigators were not able to detect significant differences in clinical outcomes over this time period. Our results serve as an updated benchmark on the usual care and outcomes of mechanically ventilated patients in a 'real-world' setting.

The investigators now propose to conduct a third international study of mechanical ventilation, 6 years after the 2nd study and 12 years after the original. This will again be a prospective, multicenter single-cohort study, which will enroll consecutive patients who have received mechanical ventilation for at least 12 hours during a 1-month period, and will follow each patient for the duration of mechanical ventilation, up to 28 days. With this 3rd study the investigators aim: 1) to determine if the observed changes that the investigators reported previously are maintained over time; 2) to evaluate if the changes implemented have impacted outcomes; 3) to analyze some aspects related to withdrawal of mechanical ventilation; and implementation non-invasive positive pressure ventilation; and 4) to evaluate what differences may occur between geographical areas.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted to the intensive care unit and require invasive mechanical ventilation (endotracheal tube or tracheostomy) for more than 12 hours.
* Patients who are admitted to the intensive care unit and require non-invasive mechanical ventilation (BIPAP or CPAP with nasal or facial mask) for more than 1 hour.

Exclusion Criteria:

* Patients less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients
Sampling Method: Probability Sample
Enrollment: 8151 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andres Esteban, MD, PhD, Study Director — Hospital Universitario de Getafe, Spain; Fernando Frutos-Vivar, MD, Principal Investigator — Hospital Universitario de Getafe, Spain; Niall D Ferguson, MD, MsC, Principal Investigator — University of Toronto, Ontario, Canada; Antonio Anzueto, MD, Principal Investigator — University of Texas Health Science Center, San Antonio, Texas, USA; Marco González, MD, Principal Investigator — Clinica Medellin & Universidad Pontificia Bolivariana, Colombia; Arnaud W Thille, MD, Principal Investigator — AP-HP, Centre Hospitalier Albert Chenevier, Henri Mondor, Créteil, France; Konstantinos Raymondos, MD, Principal Investigator — Hannover Medical School; Salvatore Maggiore, MD, Principal Investigator — Agostino Gemelli University Hospital, Università Cattolica del Sacro Cuore, Rome, Italy; Yaseen Arabi, MD, Principal Investigator — King Saud Bin Abdulaziz University for Health Sciences, Riyadh, Saudi Arabia; Rui Moreno, MD, Principal Investigator — Hospital de Santo António dos Capuchos, Lisboa, Portugal; Fekri Abroug, MD, Principal Investigator — Fattouma Bourguiba, Monastir, Tunisia; Javier Hurtado, MD, Principal Investigator — Hospital de Clínicas, Montevideo, Uruguay; Fernando Rios, MD, Principal Investigator — Hospital A.Posadas, Buenos Aires, Argentina; Luis Soto, MD, Principal Investigator — Hospital Nacional del Tórax, Santiago, Chile; Damian Violi, MD, Principal Investigator — Hospital HIGA, Güemes, Argentina; Jasmine Board, MD, Principal Investigator — Alfred Hospital, Melbourne, Australia; Andrew Davies, MD, Principal Investigator — Alfred Hospital, Melbourne, Australia; Fredi Sandi Lora, MD, Principal Investigator — Hospital Obrero Número 1, La Paz, Bolivia; Marco Antonio Soares Reis, MD, Principal Investigator — Hospital Universitário São José, Belo Horizonte, Brazil; Bin Du, MD, Principal Investigator — Peking Union Medical College Hospital, Beijing, Popular Republic of China; Hans-Henrik Bülow, MD, Principal Investigator — Holbak, Denmark; Manuel Jibaja, MD, Principal Investigator — Hospital Militar de Quito, Ecuador; Dimitros Matamis, MD, Principal Investigator — Papageorgiou Hospital, Thessaloniki, Greece; Younsuck Koh, MD, Principal Investigator — Asan Medical Center, University of Ulsan, Seoul, Korea; Asisclo Villagómez, MD, Principal Investigator — Hospital Regional 1° de Octubre, ISSSTE, México DF, Mexico; Amine Ali Zeggwagh, MD, Principal Investigator — Hôpital Ibn Sina, Rabat, Morocco; Michael Kuiper, MD, Principal Investigator — Medical Center Leeuwarden (MCL), Leeuwarden, The Netherlands; Edward Nicolayenko, MD, Principal Investigator — Hospital No.1, Moscow, Russian Federation; Nicolas Nin, MD, Principal Investigator — Hospital Universitario de Getafe, Spain; Nahit Cakar, MD, Principal Investigator — Istanbul Medical Faculty, Istanbul, Turkey; Gabriel D'Empaire, MD, Principal Investigator — Hospital de Clinicas de Caracas, Venezuela
Locations (477):
- United States (18):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville School of Medicine, Louisville, Kentucky
  - Boston Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Hospital Detroit, Detroit, Michigan
  - Omaha VA Medical Center, Omaha, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - UMDNJ-New Jersey Medical School, Newark, New Jersey
  - The Mount Sinai Medical Center, New York, New York
  - Bronx Lebanon Hospital Center, New York, New York
  - New York Methodist Hospital, New York, New York
  - Oklahoma City VA Medical Center, Oklahoma City, Oklahoma
  - Oklahoma University Health Science Center & VA medical Center, Oklahoma City, Oklahoma
  - Vanderbilt University School Of Medicine, Nashville, Tennessee
  - University Of Texas Medical Branch at Galveston, Galveston, Texas
  - University Hospital San Antonio and South Texas Veterans Health Care System, San Antonio, Texas
  - Temple Clinic, Scott & White Healthcare, Temple, Texas
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Argentina (40):
  - Hospital Naval Puerto Belgrano, Bahía Blanca
  - Clinica Bazterrica, Buenos Aires
  - Clínica Santa Isabel, Buenos Aires
  - Hospital A. Posadas, Buenos Aires
  - Hospital Churruca-Visca, Buenos Aires
  - Hospital Español, Buenos Aires
  - Hospital General de Agudos Bernardino Rivadavia, Buenos Aires
  - Hospital General de Agudos Dalmacio Vélez Sársfield, Buenos Aires
  - Hospital General de Agudos donación Francisco Santojanni, Buenos Aires
  - Hospital General de Agudos Juan A. Fernandez, Buenos Aires
  - Hospital General de Agudos P. Piñeiro, Buenos Aires
  - Hospital Municipal Coronel Suárez, Buenos Aires
  - Hospital Universitario, Universidad Abierta Interamericana, Buenos Aires
  - Sanatorio Anchorena, Buenos Aires
  - Sanatorio de la Trinidad, Buenos Aires
  - Sanatorio de los Arcos, Buenos Aires
  - Sanatorio Dr. Julio Méndez, Buenos Aires
  - Sanatorio Mater Dei, Buenos Aires
  - Sanatorio Otamendi y Miroli, Buenos Aires
  - Hospital Regional de Comodoro Rivadavia, Comodoro Rivadavia
  - Hospital Tránsito Cáceres de Allende, Córdoba
  - Sanatorio Allende, Córdoba
  - Hospital Zonal Francisco López Lima, General Roca
  - Hospital Interzonal General de Agudo Profesor Dr .Luis Guemes, Haedo
  - Hospital Interzonal de Agudos San Martin, La Plata
  - Hospital Privado de Comunidad, Mar del Plata
  - Hospital Central, Mendoza
  - Hospital Lagomaggiore, Mendoza
  - Hospital Universitario Austral, Pilar
  - Policlínico Atlántico del Sur, Río Gallegos
  - Hospital Regional Rio Grande, Río Grande
  - Hospital Provincial del Centenario, Rosario
  - Sanatorio de la Trinidad, San Isidro
  - Sanatorio Las Lomas, San Isidro
  - Hospital de San Luis, San Luis
  - Hospital Pablo Soria, San Salvador de Jujuy
  - Sanatorio Nuestra Señora del Rosario, San Salvador de Jujuy
  - Sanatorio Juncal, Temperley
  - Clínica Olivos, Vicente López
  - Clínica Privada de Especialidades de Villa María, Villa María
- Australia (20):
  - Calvary Wakefield Hospital, Adelaide
  - Flinders Medical Center, Adelaide
  - Ballarat Health Services, Ballarat
  - Bendigo Hospital, Bendigo
  - Mater Health Services, Brisbane
  - Canberra Hospital, Canberra
  - Royal Darwin Hospital, Darwin
  - Barwon Health, Geelong Hospital, Geelong
  - Royal Hobart Hospital, Hobart
  - Liverpool Hospital, Liverpool
  - Alfred Hospital, Melbourne
  - Royal Melbourne Hospital, Melbourne
  - St Vincent's Hospital, Melbourne
  - The Northern Hospital, Melbourne
  - The Western Hospital, Melbourne
  - Central Gippsland Hospital, Sale
  - Concord Hospital, Sydney
  - Nepean Hospital, Sydney
  - St George Hospital, Sydney
  - St Vincent's Hospital, Sydney
- Bolivia (2):
  - Hospital Obrero No.1, La Paz
  - Instituto Gastroenterológico, La Paz
- Brazil (23):
  - Hospital da Baleia, Belo Horizonte
  - Hospital da Polícia Militar, Belo Horizonte
  - Hospital de Pronto Socorro Risoleta Tolentino Neves, Belo Horizonte
  - Hospital Dia e Maternidade Unimed-BH, Belo Horizonte
  - Hospital Felício Rocho, Belo Horizonte
  - Hospital Júlia Kubitschek, Belo Horizonte
  - Hospital Luxemburgo, Belo Horizonte
  - Hospital Madre Teresa, Belo Horizonte
  - Hospital Nossa Senhora Aparecida, Belo Horizonte
  - Hospital São Francisco-Setimig, Belo Horizonte
  - Hospital Universitario Sao Jose, Belo Horizonte
  - Hospital Vera Cruz, Belo Horizonte
  - Hospital Vila da Serra, Belo Horizonte
  - Hospital Santa Rita, Contagem
  - Hospital São João de Deus, Divinópolis
  - Hospital de Messejana, Fortaleza
  - Hospital Universitário Walter Cantídio, Fortaleza
  - Hospital Universitário da Universidade Federal de Juiz de Fora, Juiz de Fora
  - Hospital Vaz Monteiro, Lavras
  - Santa Casa de Misericórdia de Ouro Preto, Ouro Preto
  - Hospital Arnaldo Gavazza Filho, Ponte Nova
  - Hospital Nossa Senhora das Graças, Sete Lagoas
  - Hospital São João Batista, Viçosa
- Canada (10):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - William Osler Health Science Centre, Brampton, Ontario
  - Saint Joseph Hospital, Hamilton, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Saint Michael´s Hospital, Toronto, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Hospital Western Division, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
- Chile (3):
  - Hospital de Copiapo, Copiapó
  - Hospital de Coquimbo, Coquimbo
  - Instituto Nacional del Tórax, Santiago
- China (42):
  - Beijing Chaoyang Hospital, Beijing
  - Beijing Hospital, Beijing
  - Beijing Huaxin Hospital, Beijing
  - Beijing TCM Hospital, Beijing
  - Beijing Tongren Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University 3rd Hospital, Beijing
  - PLA 304 Hospital, Beijing
  - PLA General Hospital, Beijing
  - PLA Navy General Hospital, Beijing
  - Sino-Japanese Friendship Hospital, Beijing
  - Jilin University 2nd Hospital, Changchun
  - Sichuan Provincial Hospital, Chengdu
  - West China Hospital, Chengdu
  - Chongqing Medical University 1st Hospital, Chongqing
  - Daping Hospital, Chongqing
  - Yunnan Chuxiong People's Hospital, Chuxiong
  - Dalian Medical University 1st Hospital, Dalian
  - Guangdong General Hospital, Guangdong
  - Sun Yet-Sen University 6th Hospital, Guangzhou
  - Hainan Medical College Hospital, Haikou
  - Hainan Provincial People's Hospital, Haikou
  - Zhejiang Haining People's Hospital, Haining
  - Zhejiang Tongde Hospital, Hangzhou
  - North District Hospital, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Prince Margaret Hospital, Hong Kong
  - Prince Of Wales Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Kunming City 3rd People's Hospital, Kunming
  - Kunming Medical College 1st Hospital, Kunming
  - Nanchang University 2nd Hospital, Nanchang
  - Southeast University Zhongda Hospital, Nanjing
  - Nantong 1st People's Hospital, Nantong
  - Hebei Medical University 4th Hospital, Shijiazhuang
  - Suzhou University 1st Hospital, Suzhou
  - Fengrun District People's Hospital, Tangshan
  - Wuhan University Zhongnan Hospital, Wuhan
  - Wuxi Municipal People's Hospital, Wuxi
  - Xi'an Jiaotong University 1st Hospital, Xi'an
  - Xuzhou Central Hospital, Xuzhou
  - Yantai Yuhuangding Hospital, Yantai
- Colombia (19):
  - Clínica General del Norte, Barranquilla
  - Clínica Fundadores, Bogotá
  - Clínica Shaio, Bogotá
  - Grupo Cimca Hospital de San José (medical ICU), Bogotá
  - Grupo Cimca Hospital de Suba, Bogotá
  - Grupo Cimca Hospital San José, Bogotá
  - Hospital Santa Clara, Bogotá
  - Fundación cardiovascular colombiana, Bucaramanga
  - Centro Medico Imbanaco, Cali
  - Clínica Fundación Valle Lili, Cali
  - Nuevo Hospital Bocagrande, Cartagena
  - Hospital Federico Lleras Acosta, Ibagué
  - Hospital San Rafael, Itagüí
  - Clinica Universitaria Bolivariana, Medellín
  - Clínica Cardiovascular, Medellín
  - Clínica Las Américas, Medellín
  - Clínica Medellín & Universidad Pontificia Bolivariana, Medellín
  - Corbic, Medellín
  - Hospital General de Medellín, Medellín
- Denmark (6):
  - Holbak, Holbæk
  - Koge, Køge
  - Nykobing Falster, Nykøbing Falster
  - Naestved, Næstved
  - Roskilde, Roskilde
  - Slagelse, Slagelse
- Ecuador (12):
  - Hospital José Carrasco Arteaga, Cuenca
  - Hospital Luis Vernaza, Guayaquil
  - Hospital San Vicente de Paul, Ibarra
  - Hospital Carlos Andrade Marín, Quito
  - Hospital de la Policía, Quito
  - Hospital de los Valles, Quito
  - Hospital de SOLCA (ICU medical surgical & ICU medical), Quito
  - Hospital Enrique Garcés, Quito
  - Hospital Eugenio Espejo, Quito
  - Hospital General de las Fuerzas Armadas, Quito
  - Hospital Metropolitano, Quito
  - Hospital Pablo Arturo Suárez, Quito
- Cairo University Hospitals, Cairo, Egypt
- France (11):
  - Hôpital d'Armentières, Armentières
  - Centre Hospitalier de Châlons en Champagne, Châlons-en-Champagne
  - CHU Henri Mondor, Créteil
  - CHU d'Angers, d'Angers
  - CHU De Grenoble, Grenoble
  - Centre Hospitalier Du Mans, Le Mans
  - Hôpital Édouard Herriot, Lyon
  - Centre Hospitalier De Montauban, Montauban
  - Centre Hospitalier De Roanne, Roanne
  - CHU Charles Nicolle, Rouen
  - Centre Hospitalier De Saint-Malo, St-Malo
- Germany (28):
  - Katholische Stiftung Marienhospital Aachen, Aachen
  - Universitaetsklinikum Aachen, Aachen
  - St. Nikolaus-Stiftshospital GmbH, Andernach
  - Klinikum Bad Salzungen GmbH, Bad Salzungen
  - Ermstalklinik Bad Urach, Bad Urach
  - Charité Universitaetsklinikum (ICU medical-surgical & ICU other), Berlin
  - Lungenklinik Heckeshorn, Berlin
  - Evangelisches Waldkrankenhaus Bad Godesberg gGmbH, Bonn
  - Universitaetsklinikum Bonn (ICU medical-surgical & ICU surgical), Bonn
  - Carl-Thiem-Klinikum Cottbus gGmbH, Cottbus
  - Evangelisches Krankenhaus Elisabethenstift gGmbH, Darmstadt
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Evangelisches Diakoniekrankenhaus, Freiburg im Breisgau
  - Universitaetsklinikum der Georg-August-Universitaet, Göttingen
  - Staedtisches Krankenhaus Martha-Maria Halle-Doelau gGmbH, Halle
  - Allgemeines Krankenhaus Harburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Vivantes Krankenhaus am Urban, Kreuzberg
  - Staedtisches Klinikum Lueneburg, Lüneburg
  - Universitaetsklinikum, Magdeburg
  - Hufeland Klinikum GmbH, Mühlhausen
  - Dietrich-Bonhoeffer Klinikum Neubrandenburg, Neubrandenburg
  - Klinikum der Universitaet Regensburg, Regensburg
  - Ermstalklinik Staedtisches Krankenhaus Sindelfingen, Sindelfingen
  - Bundeswehrkrankenhaus Ulm, Ulm
  - Universitaetsklinikum der Martin-Luther-Universitaet Halle-Wittenberg, Wittenberg
  - Staedtisches Klinikum Wolfenbuttel, Wolfenbüttel
  - Georgius-Agricola-Klinikum Zeitz, Zeitz
- Greece (4):
  - Agios Pavlos General Hospital, Thessaloniki
  - Ahepa Hospital, Thessaloniki
  - Gennimata Hospital, Thessaloniki
  - Papageorgiou Hospital, Thessaloniki
- Hungary (2):
  - Kenezy Hospital, Debrecen
  - University of Szeged (Four ICU), Szeged
- India (16):
  - Kalinga Hospital, Bhubaneswar
  - Apollo Hospitals, Chennai
  - Artemis Health Institute, Gūrgaon
  - CHL Apollo Hospital, Indore
  - Tata Main Hospital, Jamshedpur
  - AMRI Hospitals Kolkata, Kolkata
  - Calcutta medical research institute (CMRI), Kolkata
  - Calcutta Medical Research Institute, Kolkata
  - Kasturba Medical College, Manipal
  - Bombay Hospital Institute of Medical Sciences, Mumbai
  - Hinduja Hospital, Mumbai
  - Saifee Hospital, Mumbai
  - Tata Memorial Hospital, Mumbai
  - Ruby Hall Clinic, Pune
  - CARE Hospitals, Surat
  - Spandan Multispeciality Hospital, Vadodara
- Italy (15):
  - Ospedale Policlinico, Università Di Bari, Bari
  - Policlinico Universitario "S. Orsola-Malpighi", Bologna
  - Ospedale "San Giovanni Di Dio", Florence
  - Ospedale "Santa Maria Annunziata", Florence
  - Fondazione IRCCS "Cà Grande" Ospedale Maggiore Policlinico, Università Di Milano, Milan
  - Ospedale "San Gerardo", Università Di Milano Bicocca, Monza
  - Ospedale "V. Monaldi", Napoli
  - Ospedale Policlinico "Federico II", Università Di Napoli, Napoli
  - Ospedale Maggiore Della Carità, Università Del Piemonte Orientale "Amedeo Avogadro", Novara
  - Ospedale "Arnas Civico, Di Cristina, Benfratelli", Palermo
  - Policlinico "P. Giaccone", Università Di Palermo, Palermo
  - Fondazione IRCCS Policlinico "S. Matteo", Università Di Pavia (ICU 1 & ICU 2), Pavia
  - Policlinico "Agostino Gemelli", Università Cattolica Del Sacro Cuore, Roma
  - Policlinico "Umberto I", Università La Sapienza, Roma
  - Ospedale "San Giovanni Battista - Molinette", Università Di Torino, Torino
- Tokyo Women's Medical University, Tokyo, Japan
- Mexico (15):
  - Centenario Hospital Miguel Hidalgo, Aguascalientes
  - Hospital Regional de Pemex, Ciudad Madero
  - Hospital General de México, Mexico City
  - Instituto Nacional De Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City
  - Hospital Mérida Yucatán, Mérida
  - Hospital Juárez de México, México DF
  - Hospital Regional 1° de Octubre, ISSSTE, México DF
  - Hospital Regional de Zona No.1 del IMSS, México DF
  - Hospital Ángeles de las Lomas, México DF
  - Instituto Nacional de Cancerología, México DF
  - Umae Hospital De Especialidades Dr. Antonio Fraga Mouret, México DF
  - Centro Médico ABC, México, DF
  - Hospital Español de México, Miguel Hidalgo
  - Hospital Universitario de Nuevo León 'Dr. Eleuterio González', Nuevo León
  - Hospital Regional de Alta Especialidad de la Mujer, Villahermosa
- Morocco (3):
  - Hôpital des Specialites, Rabat
  - Hôpital Ibn Sina (Three units), Rabat
  - Hôpital Militaire D'Instruction Mohamed V, Rabat
- Netherlands (8):
  - Onze Lieve Vrouwe Gasthuis (OLVG), Amsterdam
  - Vrije Universiteit Medisch Centrum (VUMC) (Three units), Amsterdam
  - Kennemer Gasthuis, Haarlem
  - Tjongerschans Ziekenhuis, Heerenveen
  - Spaarneziekenhuis, Hoofddorp
  - Medical Center Leeuwarden (MCL), Leeuwarden
  - Universitair Medisch Centrum Maastricht, Maastricht
  - Medisch Centrum Haaglanden, The Hague
- New Zealand (7):
  - CVICU Auckland City Hospital, Auckland
  - DCCM Auckland City Hospital, Auckland
  - Middlemore, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato, Hamilton
  - Tauranga Hospital, Tauranga
  - Wellington Hospital, Wellington
- Hospital Rafael Hernández, Chiriquí, Panama
- Peru (2):
  - Hospital Edgardo Rebagliatti Martins, Lima
  - Hospital Guillermo Almenara Irigoyen, Lima
- Karol Marcinkowski University Of Medical Sciences, Poznan, Poland
- Portugal (10):
  - Hospital Garcia de Orta, Almada
  - Hospital da Luz, Amadora
  - Hospital de Cascais, Cascais
  - Centro Hospitalar de Lisboa Central, Lisbon
  - Centro Hospitalar de Lisboa Norte, Lisbon
  - Hospital de Santo Antonio dos Capuchos, Centro Hospitalar de Lisboa Central, E.P.E., Lisbon
  - Centro Hospitalar Do Porto - Hospital Geral De Santo António, Porto
  - Instituto Português de Oncología Francisco Gentil, Porto
  - Hospital De São Sebastião, Seide
  - Centro Hospitalar Trás-Os-Montes E Alto Douro, Vila Real
- VA Caribbean Health Care System, San Juan, PR, Puerto Rico
- Russia (4):
  - City Hospital Number 1 of Arkhangelsk, Arkhangelsk
  - Hospital No.7, Moscow
  - National Institute Of Surgery Named After A.V. Vishnevskij, Moscow
  - Hospital No.14, Yekaterinburg
- King Saud Bin Abdulaziz University for Health Sciences, Riyadh, Saudi Arabia
- South Korea (12):
  - Hospital Korea University of Ansan, Ansan
  - Hallym University Medical Center, Anyang
  - Hospital Chungbuk National University, Cheongju-si
  - Hospital Chuncheon Sacred Heart Hospital, Hallym University Medical Center, Chuncheon
  - Hospital Catholic University of Daegu, Daegu
  - Hospital Dongguk University of Gyeongju, Gyeongju
  - Asan Medical Center, University of Ulsan, Seoul
  - Hospital Ewha Womans University Mokdong, Seoul
  - Hospital Severance, Yonsei University Health System, Seoul
  - Samsung Medical Center, Sungkyunkwan University, Seoul
  - Hospital Yonsei University Wonju Christian, Wŏnju
  - Hospital Pusan National University of Yangsan, Yangsan
- Spain (98):
  - Hospital Juan Canalejo, A Coruña
  - Hospital General de Albacete, Albacete
  - Hospital Príncipe de Asturias, Alcalá de Henares
  - Fundación Hospital Universitario de Alcorcón, Alcorcón
  - Hospital General de Alicante, Alicante
  - Hospital San Juan, Alicante
  - Hospital Torrecárdenas, Almería
  - Hospital del Tajo, Aranjuez
  - Hospital del Sureste, Arganda
  - Hospital San Agustín, Avilés
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital de Cruces, Barakaldo
  - Hospital Clinic-IDIBAPS (ICU medical & ICU respiratory), Barcelona
  - Hospital de la Santa Creu y Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Sagrado Corazón, Barcelona
  - Hospital SCIAS, Barcelona
  - Hospital Santa María del Rosell, Cartagena
  - Hospital de la Plana, Castellon
  - Hospital General de Castellón, Castellon
  - Hospital Provincial de Castellón, Castellon
  - Hospital San Pedro de Alcántara, Cáceres
  - Complejo Hospitalario de Ciudad Real, Ciudad Real
  - Hospital del Henares, Coslada
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital de Don Benito, Don Benito
  - Complejo Hospitalario de Donostia, Donostia / San Sebastian
  - Hospital del Poniente, El Ejido
  - Hospital General Universitario de Elche, Elche
  - Hospital Arquitecto Marcide, Ferrol
  - Hospital de Fuenlabrada, Fuenlabrada
  - Hospital de Galdakao, Galdakao
  - Hospital Universitario de Getafe, Getafe
  - Hospital de Cabueñes, Gijón
  - Hospital Universitario Doctor Josep Trueta, Girona
  - Hospital Virgen de las Nieves, Granada
  - Hospital General de Guadalajara, Guadalajara
  - Hospital Juan Ramón Jimenez, Huelva
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital General de Jerez de la Frontera, Jérez de La Frontera
  - Hospital General de La Palma, La Palma
  - Hospital Doctor Negrín, Las Palmas
  - Hospital Insular de Gran Canaria, Las Palmas
  - Complejo Hospitalario de León, León
  - Hospital Arnau de Vilanova, Lleida
  - Hospital de San Pedro, Logroño
  - Complejo Hospitalario Xeral-Calde, Lugo
  - Fundación Jiménez Díaz, Madrid
  - Hospital 12 de Octubre (Trauma ICU), Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital de la Princesa, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital Quirón, Madrid
  - Hospital Universitario de la Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital de Mataró, Mataró
  - Hospital Carlos Haya, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital de Móstoles, Móstoles
  - Hospital J .M. Morales Meseguer, Murcia
  - Hospital Universitario Reina Sofia, Murcia
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Vega Baja de Orihuela, Orihuela
  - Complejo Hospitalario de Ourense, Ourense
  - Hospital Central de Asturias, Oviedo
  - Hospital Rio Carrión, Palencia
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitario Son Espasses, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Infanta Cristina, Parla
  - Complejo Hospitalario Montecelo, Pontevedra
  - Hospital Universitario de San Juan, Reus
  - Hospital Parc Taulí, Sabadell
  - Hospital de Sagunto, Sagunto
  - Complejo Hospitalario de Salamanca, Salamanca
  - Hospital Clínico de Salamanca, Salamanca
  - Complejo Hospitalario de Santiago de Compostela, Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - Hospital Universitario de Valme, Seville
  - Hospital Virgen del Rocío, Seville
  - Hospital General de Soria, Soria
  - Hospital Mutua de Terrassa, Terrassa
  - Hospital Obispo Polanco, Teruel
  - Complejo Hospitalario de Toledo, Toledo
  - Hospital de Torrevieja, Torrevieja
  - Hospital Infanta Elena, Valdemoro
  - Hospital Universitario de la Fe, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Clínico de Valladolid, Valladolid
  - Hospital Rio Hortega, Valladolid
  - Hospital Meixoeiro, Vigo
  - Hospital Santiago Apóstol, Vitoria-Gasteiz
  - Hospital Lluis Alcanyis, Xàtiva
  - Hospital de Zamora, Zamora
  - Hospital Clínico Lozano Blesa, Zaragoza
  - Hospital Royo Vilanova, Zaragoza
- Chi Mei Medical Center, Tainan, Taiwan
- Tunisia (5):
  - Hospital Abderrahmane Mami, Aryanah
  - Hospital Taher Sfar City, Mahdia
  - Hospital Fattouma Bourguina (ICU medical & ICU surgical), Monastir
  - CHU Habib Bourguiba, Sfax
  - Hospital Universitarie Farhat Hached, Sousse
- Turkey (Türkiye) (8):
  - Uludag University Faculty of Medicine, Bursa
  - Erciye Üniversity, Erciyes
  - Anadolu Medical Center Istanbul, Istanbul
  - Atatürk Hospital, Izmir
  - Sutcu İmam University, Kahramanmaraş
  - Kirikkale University, Kırıkkale
  - Faculty of Medicine Mersin University, Mersin
  - Medical Faculty of Yuzuncu Yil University, Van
- Uruguay (22):
  - CAAMOC Carmelo, Carmelo
  - Orameco, Colonia del Sacramento
  - Hospital de Florida, Florida
  - CRAMI, Las Piedras
  - Hospital de Maldonado, Maldonado
  - Sanatorio Mautone, Maldonado
  - Sanatorio CAMS, Mercedes
  - CASMU Nº2, Montevideo
  - Circulo Católico, Montevideo
  - CUDAM, Montevideo
  - Hospital de Clínicas, Montevideo
  - Hospital Español, Montevideo
  - Hospital Evangélico, Montevideo
  - Hospital Maciel, Montevideo
  - Hospital Pasteur, Montevideo
  - Hospital Policial, Montevideo
  - Impassa, Montevideo
  - Sanatorio Americano, Montevideo
  - CAAMEPA, Pando
  - COMEPA, Paysandú
  - Hospital Escuela del Litoral, Paysandú
  - Sanatorio Cantegril, Punta del Este
- Venezuela (4):
  - Hospital Centro de Especialidades, Anzoátegui
  - Hospital Clínico Universitario, Caracas
  - Hospital de Clínicas, Caracas
  - Hospital Miguel Pérez Carreño, Caracas
- Viet Duc Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Esteban A, Anzueto A, Frutos F, Alia I, Brochard L, Stewart TE, Benito S, Epstein SK, Apezteguia C, Nightingale P, Arroliga AC, Tobin MJ; Mechanical Ventilation International Study Group. Characteristics and outcomes in adult patients receiving mechanical ventilation: a 28-day international study. JAMA. 2002 Jan 16;287(3):345-55. doi: 10.1001/jama.287.3.345. PMID 11790214
- [Background] Esteban A, Ferguson ND, Meade MO, Frutos-Vivar F, Apezteguia C, Brochard L, Raymondos K, Nin N, Hurtado J, Tomicic V, Gonzalez M, Elizalde J, Nightingale P, Abroug F, Pelosi P, Arabi Y, Moreno R, Jibaja M, D'Empaire G, Sandi F, Matamis D, Montanez AM, Anzueto A; VENTILA Group. Evolution of mechanical ventilation in response to clinical research. Am J Respir Crit Care Med. 2008 Jan 15;177(2):170-7. doi: 10.1164/rccm.200706-893OC. Epub 2007 Oct 25. PMID 17962636
- [Derived] Nin N, Muriel A, Penuelas O, Brochard L, Lorente JA, Ferguson ND, Raymondos K, Rios F, Violi DA, Thille AW, Gonzalez M, Villagomez AJ, Hurtado J, Davies AR, Du B, Maggiore SM, Soto L, D'Empaire G, Matamis D, Abroug F, Moreno RP, Soares MA, Arabi Y, Sandi F, Jibaja M, Amin P, Koh Y, Kuiper MA, Bulow HH, Zeggwagh AA, Anzueto A, Sznajder JI, Esteban A; VENTILA Group. Severe hypercapnia and outcome of mechanically ventilated patients with moderate or severe acute respiratory distress syndrome. Intensive Care Med. 2017 Feb;43(2):200-208. doi: 10.1007/s00134-016-4611-1. Epub 2017 Jan 20. PMID 28108768
- [Derived] Esteban A, Frutos-Vivar F, Muriel A, Ferguson ND, Penuelas O, Abraira V, Raymondos K, Rios F, Nin N, Apezteguia C, Violi DA, Thille AW, Brochard L, Gonzalez M, Villagomez AJ, Hurtado J, Davies AR, Du B, Maggiore SM, Pelosi P, Soto L, Tomicic V, D'Empaire G, Matamis D, Abroug F, Moreno RP, Soares MA, Arabi Y, Sandi F, Jibaja M, Amin P, Koh Y, Kuiper MA, Bulow HH, Zeggwagh AA, Anzueto A. Evolution of mortality over time in patients receiving mechanical ventilation. Am J Respir Crit Care Med. 2013 Jul 15;188(2):220-30. doi: 10.1164/rccm.201212-2169OC. PMID 23631814

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive patients who required mechanical ventilation for more than 12 hours in the participating intensive care units.
Period: Overall Study
Arm/Group | Mechanically Ventilated Patients
Started | 8151
Completed | 8151
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mechanically Ventilated Patients
Number analyzed (Participants) | 8151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4233
  >=65 years | 3918
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3105
  Male | 5046

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Description: Mortality at discharge from intensive care unit
Time Frame: At day 28 after the beginning of mechanical ventilation
Measure: Count of Participants; unit: Participants
Arm/Group | Mechanically Ventilated Patients
Number analyzed (Participants) | 8151
Participants | 2269

ADVERSE EVENTS:
Arm/Group | Mechanically Ventilated Patients
All-Cause Mortality (participants affected / at risk) | 2269/8151
Serious Adverse Events (participants affected / at risk) | 0/8151
Other Adverse Events (participants affected / at risk) | 0/8151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No